CLINICAL TRIAL: NCT05855252
Title: PRECISION-TBI - A Multi-centre Prospective Observational Cohort Study of Patients With Moderate to Severe Traumatic Brain Injury
Brief Title: PRECISION-TBI - An Observational Study of Patients With Moderate to Severe Traumatic Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: ANZIC-RC/AU001
Record Dates: First submitted 2023-03-28; First posted 2023-05-11 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Trauma, Brain
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Traumatic Brain Injury (TBI) is a devastating condition and a leading cause of long-term disability. Every patient with TBI has a different type of injury and is treated differently from hospital to hospital making it very difficult to identify the most effective treatments. The current study focuses on the most severe types of TBI that require hospital ICU care - moderate to severe TBI (m-sTBI). The overall aim of this study is to collect data about how different hospitals manage m-sTBI in Australia, and to quantify the variability that likely exists. Recovery at 6 months post-injury will be collected to allow a better understanding on how different injuries and treatments affect long term outcomes.

DETAILED DESCRIPTION:
Traumatic Brain Injury (TBI) is a devastating condition and a leading cause of death and long-term disability, particularly in young adults. In Australia and New Zealand, severe TBI accounts for over 700 intensive care unit (ICU) admissions per year. Approximately half of these patients will die or be severely disabled six months after their injury. The lifetime costs for the disabled survivors of TBI reach an estimated $1 billion annually. There are strong ethical, medical, social and health economic reasons to improve treatment and reduce disability in TBI.

TBI is a broad term for many different types of injuries to the brain. This study focuses on the most severe types of TBI that require hospital management and ICU care - moderate to severe TBI (m-sTBI). The fact that every patient with m-sTBI is different, has a different type of injury and is treated differently from hospital to hospital makes it very difficult to study m-sTBI and identify the most effective treatments for improving patient outcomes. At the moment, there is only a small amount of data on how m-sTBI patients are treated in the different hospitals in Australia and whether there are differences in outcomes associated with different approaches to m-sTBI management. Currently there is no central database for m-sTBI patients in Australia that can be used to compare different hospitals and track progress over time.

The first aim of PRECISION-TBI is to collect data about how different hospitals manage m-sTBI in Australia, and to quantify the variability that likely exists. High quality data about the initial injury (cause, severity and presence of factors that may make the injury worse), the early management of the patient (e.g. time to arrival at hospital), the surgical management of the patient (surgeries undertaken and monitoring probes utilised), the clinical management in ICU and neurological outcome after the injury will be collected. The main focus will be on the ICU management of m-sTBI so participating sites will be provided with computers and specialist software to collect accurate minute to minute data from brain monitors used to guide patient management in the ICU. Recovery at 6 months post-injury will be collected for all enrolled participants to understand how different injuries and treatments have affected long term patient outcomes.

The participating hospitals will also be provided with feedback on the characteristics of their m-sTBI patient population, the treatments that they are using and the outcomes for their patients. It will be possible for participating hospitals to compare each of these parameters with other similar hospitals and this will allow the identification of any factors that are strongly associated with improved patient outcomes. This will be provided over the course of at least 2 years, which will allow hospitals to track progress over time and identify how changes to management protocols and care systems may result in better outcomes for patients in this highly vulnerable group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosis of moderate to severe TBI
* Insertion of invasive intra-cranial monitoring
* Study inclusion within 48 hours of ICU admission

Exclusion Criteria:

* Admission to the ICU is solely for the purposes of palliative care or confirmation of organ donation
* Advanced care directive or previously stated wish not to be included in research activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: moderate to severe traumatic brain injured patients who are admitted to the intensive care unit.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-14 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Glasgow outcome scale | At 6 months post-injury
  Unfavourable outcome at 6 months post-injury (defined as a score of 4 or less on the 8-point extended Glasgow outcome scale)

SECONDARY OUTCOMES:
Mortality | Up to 6 months post-injury
  Death occurring any time between date of hospital admission and 6 months post-injury (up to 180 days post-injury)
Hospital length of stay | Through study completion, an average of 1 year
  Number of acute hospital admission days
Intensive care Unit (ICU) length of stay | Through study completion, an average of 1 year
  Number of ICU admission days
EuroQol (EQ-5D five-level) | At 6 months post-injury
  Quality of life questionnaire, each of the 5 questions is scored from 1 (no problem performing that particular task) to 5 (unable to perform the task).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Udy, MB,FCICM,PhD, Principal Investigator — Monash University
Locations (9):
- Australia (9):
  - St George Hospital, Kogarah, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeffcote T, Battistuzzo CR, Plummer MP, McNamara R, Anstey J, Bellapart J, Roach R, Chow A, Westerlund T, Delaney A, Bihari S, Bowen D, Weeden M, Trapani A, Reade M, Jeffree RL, Fitzgerald M, Gabbe BJ, O'Brien TJ, Nichol AD, Cooper DJ, Bellomo R, Udy A. PRECISION-TBI: a study protocol for a vanguard prospective cohort study to enhance understanding and management of moderate to severe traumatic brain injury in Australia. BMJ Open. 2024 Feb 21;14(2):e080614. doi: 10.1136/bmjopen-2023-080614. PMID 38387978